CLINICAL TRIAL: NCT06966362
Title: Varenicline for Smoking Reduction in Veterans Unwilling to Quit
Brief Title: Varenicline for Smoking Reduction in Veterans Not Ready To Quit
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NURA-007-24F
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Veterans; Tobacco Use Disorder; Cigarette Smoking; Tobacco Dependence
Keywords: Varenicline; Tobacco use disorder; Veterans; Quit attempts; Cigarette smoking; Motivation phase treatment; Nicotine replacement therapy; Smoking reduction; Smoking abstinence
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking; Smoking Reduction | interventions — Varenicline; Nicotine Chewing Gum; Nicotine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two 12-week Motivation-phase treatment groups: (1) varenicline, or (2) NRT (2 mg mini-lozenges).
Who Masked: Outcomes Assessor
Masking Description: Only the outcome assessors will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motivation-Phase Varenicline (Experimental): Varenicline use during pre-quit phase of smoking treatment for participants who are interested in cutting down on their smoking.
  Interventions: Drug: Motivation-Phase Varenicline; Drug: Cessation-Phase Varenicline; Behavioral: Motivation-Phase Counseling; Behavioral: Cessation-Phase Counseling
- Motivation-Phase Nicotine Mini-Lozenge (Active Comparator): NRT mini-lozenge use during pre-quit phase of smoking treatment for participants who are interested in cutting down on their smoking.
  Interventions: Drug: Motivation-Phase Nicotine Mini-Lozenge; Drug: Cessation-Phase Combination Nicotine Replacement Therapy (NRT); Behavioral: Motivation-Phase Counseling; Behavioral: Cessation-Phase Counseling

INTERVENTIONS:
Drug: Motivation-Phase Varenicline — Varenicline reduction dosing will start when participants initiate Motivation-phase treatment: 0.5mg once daily for 3 days, increasing to 0.5mg twice daily for days 4 to 7, and then to the maintenance dose of 1mg twice daily for the duration of the 12-week reduction regimen.
  Other Names: Chantix
  Arms: Motivation-Phase Varenicline
Drug: Motivation-Phase Nicotine Mini-Lozenge — NRT mini-lozenge reduction dosing will start when participants initiate Motivation-phase treatment: 2-mg mini-lozenges in place of cigarettes (5-15/day).
  Other Names: Nicorette
  Arms: Motivation-Phase Nicotine Mini-Lozenge
Drug: Cessation-Phase Combination Nicotine Replacement Therapy (NRT) — Combination NRT (nicotine patch + nicotine mini-lozenge) cessation dosing will begin on the target quit day: if smoking >10 cigarettes/day = 8 weeks of 21-mg, 2 weeks of 14-mg, and 2 weeks of 7-mg nicotine patches; if smoking 10 cigarettes/day = 10 weeks of 14-mg and 2 weeks of 7-mg nicotine patches. All participants will receive 2 or 4 mg mini-lozenge for the 12-week cessation period (9/day, 1 piece every 1-2/hours).
  Other Names: Nicorette, Nicoderm
  Arms: Motivation-Phase Nicotine Mini-Lozenge
Drug: Cessation-Phase Varenicline — Varenicline cessation dosing will start one week prior to their TQD: 0.5mg once daily for 3 days, increasing to 0.5mg twice daily for days 4 to 7, and then to the maintenance dose of 1mg twice daily for the remainder of the 12-week cessation regimen.
  Other Names: Chantix
  Arms: Motivation-Phase Varenicline
Behavioral: Motivation-Phase Counseling — All participants receive motivation-phase counseling. Motivation-phase counseling involves 5, 10-15-minute counseling calls. The counselor will work with participants on smoking control skills selected by the participant, such as avoidance of smoking cues, reducing smoking heaviness/contexts, developing urge coping skills, or finding support from friends and family. Counseling will emphasize setting realistic and achievable smoking control goals. Counseling will also emphasize competence and self-efficacy, which will be linked to success in smoking control.
Behavioral: Cessation-Phase Counseling — All participants who enter cessation treatment will be offered 4, 10-15-minute counseling calls. The first counseling session involves pre-quit preparation, and can occur any time before the target quit day. The other 3 counseling calls will be scheduled for 1 day, 1 week, and 4 weeks after the target quit date. Cessation counseling will be based on treatment guidelines and will review instructions for when to start cessation medication, the timing of the quit day (relative to medication start), and medication adherence. Counseling will involve problem solving and skill development.

SUMMARY:
In order to reduce the prevalence of cigarette smoking among Veterans, it is vital that healthcare providers offer effective tobacco treatment to all Veterans who smoke, including those not ready to make a quit attempt. Smoking treatments currently available to Veterans who are not ready to quit are only weakly effective. This project will generate new knowledge about the effectiveness of a promising varenicline-based intervention designed to increase quit attempts and long-term abstinence in Veterans who are initially not ready to quit. This project has great potential to engage Veterans not ready to quit smoking in treatment that increases quit attempts and quitting success, thereby reducing morbidity and mortality caused by smoking in Veterans.

DETAILED DESCRIPTION:
Evidence-based smoking cessation treatments can double smoking abstinence rates, yet these treatments are underused by the millions of Veterans who smoke. One reason for this is that the great majority of people who smoke are not ready to make a quit attempt when cessation treatment is offered (70-90%). An important public health goal is to increase engagement of people not ready to quit smoking in highly effective treatment that prepares them to make quit attempts and ultimately achieve abstinence (i.e., Motivation-phase treatment; MPT). MPT typically combines smoking reduction counseling with nicotine replacement therapy (NRT). Although offering NRT Motivation-phase treatment (NRT MPT) in healthcare settings increases the reach of tobacco treatment, such interventions only weakly affect long-term abstinence. It is vital that the investigators develop more effective MPTs that increase quit attempts and quitting success in people not ready to quit. Varenicline, the most effective single agent smoking cessation pharmacotherapy, holds great promise as an intervention for people who are not ready to make a quit attempt. The investigators propose that MPT will be markedly more effective if it involves the use of varenicline (vs. NRT) because it will more effectively reduce smoking reward, affective withdrawal, and tonic craving. Initial evidence suggests that varenicline increases quitting motivation in those not ready to quit, but the extant studies have not 1) directly evaluated varenicline effectiveness in this population and 2) compared varenicline MPT with NRT MPT, the current standard treatment for those not ready to make a quit attempt. The goal of this study is to evaluate whether varenicline MPT is especially effective and cost-effective relative to NRT MPT, in Veterans who are willing to reduce but not quit smoking. This study will compare the use of varenicline MPT vs. NRT MPT on: biochemically verified point-prevalence abstinence at 1 year (primary outcome), quit attempts, and cessation treatment use.

This study is a 2-group randomized controlled trial that will enroll 400 adults from three geographically diverse VA hospitals who smoke 5 cigarettes/day and do not want to quit smoking in the next 30 days but are willing to cut down. Participants will be randomized to one of two 12-week MPT groups: (1) varenicline, or (2) NRT (2 mg mini-lozenges). All participants will receive 5 phone counseling sessions focused on smoking reduction during the 12-week MPT. Any participants who decide to try quitting will receive smoking cessation treatment involving continued use of their assigned study medication and cessation counseling.

ELIGIBILITY:
Inclusion Criteria:

* Report smoking an average of 5 or more cigarettes daily for the previous 6 months
* Not ready to set a quit date in the next 30 days but willing to cut down on their smoking
* Able to read, write, and speak English
* Be medically eligible to use study medications (NRT or varenicline)
* If female, use an approved method of birth control while using study medication
* Be at least 21 years old
* Be a Veteran

Exclusion Criteria:

* Unable to give informed, voluntary consent to participate
* Current use of any pharmacotherapy for smoking cessation
* Use of non-cigarette tobacco products as primary form of tobacco use
* Incarceration

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2031-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Biochemically confirmed 7-day point-prevalence abstinence | 12 months post-study entry
  Participants who report 7-day point-prevalence abstinence from cigarettes at the 12 month follow-up will mailed a saliva collection kit that will test cotinine and anabasine to validate self-reported abstinence from combusted tobacco.

SECONDARY OUTCOMES:
7-day point prevalence abstinence | 6 months post-study entry
  Participants who report 7-day point-prevalence abstinence from cigarettes at the 6 month follow-up will mailed a saliva collection kit that will test cotinine and anabasine to validate self-reported abstinence from combusted tobacco.
Making a quit attempt lasting 24 hours | 6 and 12 months post-study entry
  Making a quit attempt lasting at least 24 hours by 6 and 12 months; coded as binary (0 or 1).
Cessation treatment entry | 6 months post-study entry
  Entering cessation treatment; coded as binary (0 or 1)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Megan Cook, PhD, Principal Investigator — William S. Middleton Memorial Veterans Hospital, Madison, WI; Neal M Doran, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (4):
- United States (4):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Deidentified dataset will be shared upon request.